CLINICAL TRIAL: NCT05816226
Title: Comparison of Topical 1% Diclofenac and Topical 2.5% Hydrocortisone for TMJ Arthralgia
Brief Title: Topical Treatment for TMJ Arthralgia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of the Pacific (Other)
Responsible Party: Principal Investigator, Andrew Young, Assistant Professor, Department of Diagnostic Sciences, University of the Pacific
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023 Young A 1
Record Dates: First submitted 2023-04-03; First posted 2023-04-18 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: TMJ Pain
Keywords: diclofenac; hydrocortisone; TMJ; arthralgia
MeSH Terms: conditions — Arthralgia | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Cream containers labeled by randomly-generated numbers, by person not involved in analysis or patient interaction.
  Statistical analysis done by person not aware of the treatment received by each group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydrocortisone topical (Experimental): 2.5% hydrocortisone cream
  Interventions: Drug: Hydrocortisone 2.5%
- Diclofenac topical (Active Comparator): 1% diclofenac cream
  Interventions: Drug: Diclofenac 1% topical

INTERVENTIONS:
Drug: Hydrocortisone 2.5% — Applied four times daily to TMJ with arthralgia
  Arms: Hydrocortisone topical
Drug: Diclofenac 1% topical — Applied four times daily to TMJ with arthralgia
  Arms: Diclofenac topical

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of topical 2.5% hydrocortisone in TMJ arthralgia. The main questions it aims to answer are:

* How does pain reduction compare?
* How does improvement in jaw function limitation compare?
* How do side effects compare? Participants will
* On day 1 be examined and report their pain level and jaw function limitation
* On days 1-21, apply their cream four times a day
* On day 21, report their pain level, jaw function limitation, compliance with instructions, and side effects.

Researchers will compare topical 2.5% hydrocortisone and topical 1% diclofenac to see if efficacy and side effects differ.

DETAILED DESCRIPTION:
* Person 2 will label creams, patient packets (pre-stamped envelope, questionnaire, consent form), and give packets to Person 1 in the order in which they are to be dispensed.
* Person 1 will recruit all eligible patients in the order in which they are seen, enrolling all that consent. Packets and gel will be given to patient, and written and verbal instructions, including that email will be sent saying "Keep it up!" to remind them to continue applying get, as well as "Please send us your questionnaire". Consent forms will be stored in locked drawer.
* Person 1 will remind patient on days 7 and 14 to continue with the study
* Person 1 will remind patient on day 21 to mail back the completed questionnaire
* Person 1 will reach out to all patients from whom the questionnaire is not returned within 1 week of day 21, and do so at weekly intervals a minimum of 3 times.
* Person 1 will enter data in Excel as it comes, reaching out to patients if there are questions. Excel file uses random number ID, not patient name, thereby anonymizing the data
* Persons 1, 2, 3, and 4 will decide which patient's data, if any, should be removed
* Person 1 will send complete anonymized Excel data file (containing all patients) to Person 3
* Person 2 will determine, using random number generator, which group will be referred to as "Group A" during the statistical analysis, and which will be referred to as "Group B"
* Person 2 will tell Dr. Korczeniewska which data will be in Group A, and which will be in Group B
* Person 3 will perform statistical analysis
* Person 2 will reveal which group was Hydrocortisone, and which was Diclofenac

ELIGIBILITY:
Inclusion Criteria:

* Arthralgia of at least 1 TMJ for at least 3 days

Exclusion Criteria:

* Systemic pain condition
* Past adverse reaction to steroid
* Currently taking steroid
* Taken steroid in the past ___ months
* Muscle relaxants (may start after study is complete)
* New night guard during study, or within 1 month of start of study (may start after study is complete)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity | Pain measured on days 1 and 21
  Using Visual Analog Scale, Range 0 - 10 cm, with 0 cm = no pain, and 10 cm = extreme pain
Change in jaw function limitation | Jaw function limitation measured on days 1 and 21
  Using jaw function limitation scale, Range 0-10 for each of the 8 parameters, with 0 = no limitation, and 10 = severe limitation

SECONDARY OUTCOMES:
Number of participants with side effects | Reported on day 21
  Write-in side effects, select intensity (mild, moderate, severe), write in length of each occurrence, and % of times it occurred with cream application

CONTACTS AND LOCATIONS:
Locations (1):
- Arthur A. Dugoni School of Dentistry, University of the Pacific, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bariguian Revel F, Fayet M, Hagen M. Topical Diclofenac, an Efficacious Treatment for Osteoarthritis: A Narrative Review. Rheumatol Ther. 2020 Jun;7(2):217-236. doi: 10.1007/s40744-020-00196-6. Epub 2020 Feb 21. PMID 32086778
- [Background] Wade AG, Crawford GM, Young D, Corson S, Brown C. Comparison of diclofenac gel, ibuprofen gel, and ibuprofen gel with levomenthol for the topical treatment of pain associated with musculoskeletal injuries. J Int Med Res. 2019 Sep;47(9):4454-4468. doi: 10.1177/0300060519859146. Epub 2019 Jul 29. PMID 31353997
- [Background] Niethard FU, Gold MS, Solomon GS, Liu JM, Unkauf M, Albrecht HH, Elkik F. Efficacy of topical diclofenac diethylamine gel in osteoarthritis of the knee. J Rheumatol. 2005 Dec;32(12):2384-92. PMID 16331769